CLINICAL TRIAL: NCT04585165
Title: Cohort of Individuals at Risk of HIV Infection Recruited in User-friendly HIV Testing and Counseling Services in Thailand Provinces
Brief Title: User-friendly HIV Testing and Counseling Services
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Expertise France-L'Initiative (Unknown); French National Research Institute for Sustainable Development (IRD) (Unknown)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, Researcher, Chiang Mai University
Other Study IDs: Napneung-2
Record Dates: First submitted 2020-04-27; First posted 2020-10-14 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: HIV Infections; Sexually Transmitted Infection; Hepatitis B, Chronic; Hepatitis C
Keywords: HIV; Testing; Self-testing; Retesting; Early diagnosis; Counseling; Computer; Reminder; Short message service; Pre-exposure prophylaxis
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Hepatitis B, Chronic; Hepatitis C; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma from remaining blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Risk of HIV acquisition: Individuals reporting behavioral risk of HIV acquisition.

SUMMARY:
Multicenter cohort study of individuals reporting behavioral risks of HIV acquisition, recruited among those presenting for testing for HIV and other sexually transmitted infections.

Overarching goal: to study factors associated with uptake of HIV prevention and (re)testing services in medium-sized cities in Thailand.

Primary objective: To estimate the incidence of HIV and other sexually transmitted infections (syphilis, chronic hepatitis B and C) among individuals presenting for retesting.

Secondary objectives:

* To evaluate the uptake of pre-exposure prophylaxis
* To assess retention in the study
* To evaluate client HIV knowledge
* To describe HIV prevalence and characteristics of individuals newly diagnosed with HIV
* To describe characteristics of individuals at risk of HIV infection
* To assess the quality of the testing and referral services.

DETAILED DESCRIPTION:
Testing and counseling for HIV, syphilis and other sexually transmitted infections is provided to consenting individuals.

Components: interactive counseling program, self sampling (finger prick) under supervision, questionnaire (on a tablet computer) to assess risks of HIV acquisition, understanding of HIV transmission routes and pre-exposure prophylaxis, willingness to take pre-exposure prophylaxis if at risk of HIV, and satisfaction with regard to services provided.

Referral to appropriate care facility of participants diagnosed with infection. HIV negative participants with significant risk of HIV are advised to come back for HIV retesting within 3 to 6 months and informed about pre-exposure prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 years or more
* Willing to be tested for HIV and other sexually transmitted infections
* Able to understand the study and its procedures

Exclusion Criteria: None

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals requesting a test for HIV and sexually transmitted infections
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
HIV incidence | Through study completion, an average of 3 years
  HIV incidence

SECONDARY OUTCOMES:
Participants initiating pre-exposure prophylaxis | Through study completion, an average of 3 years
  Proportion of participants initiating pre-exposure prophylaxis among those at significant risk of HIV
Retention | Through study completion, an average of 3 years
  Cumulative probability of retest
HIV knowledge | Through study completion, an average of 3 years
  Answers to a self-constructed questionnaire assessing participants' knowledge of HIV transmission routes and pre-exposure prophylaxis, following counseling. The questionnaire is composed of one multiple-choice question on HIV transmission routes and three True/False questions on pre-exposure prophylaxis. The results will be reported item by item. Exploratory data analyses may be conducted using, for example, principal component analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzague Jourdain, MD, PhD, Principal Investigator — Chiang Mai University
Locations (6):
- Thailand (6):
  - STIs Clinic of the Office of Disease Prevention and Control Region 1, Chiang Mai
  - Clinical Service Center, Faculty of Associated Medical Sciences, Chiang Mai University, Chiang Mai
  - MAP Foundation, Chiang Mai
  - Chiang Rai Obstetrics Clinic, Chiang Rai
  - Phayao Hospital, Phayao
  - University of Phayao Medical Center and Hospital, Phayao

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salvadori N, Decker L, Ngo-Giang-Huong N, Mary JY, Chevret S, Arunothong S, Adam P, Khamduang W, Samleerat T, Luangsook P, Suksa-Ardphasu V, Achalapong J, Rouzioux C, Sirirungsi W, Jourdain G. Impact of Counseling Methods on HIV Retesting Uptake in At-Risk Individuals: A Randomized Controlled Study. AIDS Behav. 2020 May;24(5):1505-1516. doi: 10.1007/s10461-019-02695-2. PMID 31605294
- [Background] Salvadori N, Adam P, Mary JY, Decker L, Sabin L, Chevret S, Arunothong S, Khamduang W, Luangsook P, Suksa-Ardphasu V, Achalapong J, Rouzioux C, Sirirungsi W, Ngo-Giang-Huong N, Jourdain G. Appointment reminders to increase uptake of HIV retesting by at-risk individuals: a randomized controlled study in Thailand. J Int AIDS Soc. 2020 Apr;23(4):e25478. doi: 10.1002/jia2.25478. PMID 32294318
- See also: Presentation for potential participants — https://www.napneung.net/